CLINICAL TRIAL: NCT07130760
Title: Is Intraligamentary Injection the Anesthesia of Choice for Symptomatic Irreversible Pulpitis in Mandibular Molars? A Multicenter Randomized Comparative Trial.
Brief Title: Intraligamentary vs Inferior Alveolar Nerve Block for Pulpitis: A Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator - DDS, PhD (Bioengineering), Aula Dental Avanzada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILA VS AINB PULP
Record Dates: First submitted 2025-06-05; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-06

CONDITIONS: Symptomatic Irreversible Pulpitis (SIP); Dental Pain; Inferior Alveolar Nerve Block Failure; Local Anesthesia
Keywords: Inferior alveolar nerve block; Pulpitis Mandibular molars; Emergency dental treatment; Symptomatic irreversible pulpitis; Randomized clinical trial; Endodontics; Dental pain; Local anesthesia; Intraligamentary anesthesia
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either intraligamentary injection or inferior alveolar nerve block prior to endodontic treatment of mandibular molars with symptomatic irreversible pulpitis.
Who Masked: Participant
Masking Description: Participants will be unaware of which anesthetic technique is administered. Operators cannot be blinded due to the nature of the procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraligamentary Injection Group (Experimental): Patients in this arm will receive intraligamentary anesthesia prior to endodontic access.
  Interventions: Procedure: Intraligamentary Injection
- Inferior Alveolar Nerve Block Group (Active Comparator): Patients in this arm will receive standard inferior alveolar nerve block prior to endodontic access.
  Interventions: Procedure: Inferior Alveolar Nerve Block

INTERVENTIONS:
Procedure: Intraligamentary Injection — Intraligamentary local anesthesia will be administered using a standard dental syringe with 2% lidocaine and 1:100,000 epinephrine.
  Other Names: Intraligamental anesthesia (ILA); Periodontal ligament injection (PDL injection); Intraligamentary anesthetic technique
  Arms: Intraligamentary Injection Group
Procedure: Inferior Alveolar Nerve Block — Inferior alveolar nerve block will be performed with 2% lidocaine and 1:100,000 epinephrine using the conventional technique.
  Other Names: Inferior alveolar nerve anesthesia; Inferior dental block
  Arms: Inferior Alveolar Nerve Block Group

SUMMARY:
This multicenter randomized trial compares the clinical effectiveness of intraligamentary injection versus inferior alveolar nerve block (IANB) in patients with symptomatic irreversible pulpitis in mandibular molars. The goal is to determine which technique provides better pain control during endodontic treatment.

DETAILED DESCRIPTION:
Symptomatic irreversible pulpitis in mandibular molars presents a clinical challenge due to the difficulty in achieving profound anesthesia. This prospective, randomized, controlled clinical trial evaluates two anesthetic techniques-intraligamentary injection (ILA) versus inferior alveolar nerve block (IANB)-to compare their efficacy in eliminating pain during endodontic access. Patients will be enrolled from multiple dental centers following standardized inclusion and exclusion criteria. Pain will be assessed using validated scales. Statistical analysis will be conducted to determine significant differences in anesthetic success between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Presenting with symptomatic irreversible pulpitis in a mandibular molar
* Vital response to cold testing
* Ability to understand and provide informed consent
* Available for follow-up and data collection

Exclusion Criteria:

* Known allergy to lidocaine or epinephrine
* Pregnancy or breastfeeding
* Use of analgesics or anti-inflammatory drugs in the previous 6 hours
* Non-vital or previously treated teeth
* Significant systemic disease (ASA III or above)
* History of psychiatric or neurological disorders affecting pain perception

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Pain during endodontic access | Immediately after access cavity preparation (within 30 minutes of anesthesia)
  Pain intensity experienced by the patient during endodontic access after the assigned anesthetic technique.

SECONDARY OUTCOMES:
Need for supplementary anesthesia | During access or initial root canal instrumentation (within first 45 minutes)
  Whether the initial anesthesia technique was sufficient or required additional anesthetic injection to complete the procedure pain-free.
Patient satisfaction immediately after treatment | End of visit (within 1 hour)
  Patient-reported satisfaction immediately after treatment will be measured using a 5-point Likert scale. The scale ranges from 1 (very dissatisfied) to 5 (very satisfied). Higher scores indicate better satisfaction.
Postoperative pain at 7 days | Day 7 post-treatment
  Pain intensity reported by the patient at day 7 after treatment will be assessed using a 4-point ordinal scale: 1 (none), 2 (mild), 3 (moderate), 4 (severe). Higher scores indicate worse pain.
Patient satisfaction at 7 days | Day 7 post-treatment
  Patient-reported satisfaction one week after treatment will be measured using a 5-point Likert scale. The scale ranges from 1 (very dissatisfied) to 5 (very satisfied). Higher scores indicate better satisfaction.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clínica Dental 4, Ferrol, A coruña
  - Clínica Dental Esteve, Alicante, Alicante

IPD SHARING:
Plan to Share IPD: No
This study will not share individual participant data (IPD).